CLINICAL TRIAL: NCT05048914
Title: Migraine Abortive Treatment in Children and Adolescents in Israel
Brief Title: Migraine Abortive Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, Jacob.genizi, Director Pediatric Neurology Unit, Bnai Zion Medical Center
Other Study IDs: BNZ 095-19
Record Dates: First submitted 2021-09-09; First posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Ibuprofen; Acetaminophen; Dipyrone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ibuprofen — treatment of acute migraine attack
  Other Names: acetaminophen; dipyrone

SUMMARY:
Migraine headaches in children and adolescents may cause severe attacks that require abortive treatment. This study evaluated the incidence and efficacy of medications used for relieving migraine headache attacks in the pediatric population in Israel. Children 6-18 years of age who were diagnosed in our pediatric neurology clinic as having migraine headaches were enrolled into the study. Children and their parents filled in questionnaires about their response to abortive treatment two hours after use, during three acute headache attacks. The questionnaire included demographic data, baseline headache intensity, migraine-associated symptoms, medications used, and pain assessment.

DETAILED DESCRIPTION:
Background: Headaches are a common complaint in children and adolescents. Most cases are caused by a benign problem or a primary headache disorder, such as migraine and tension-type headaches. Not enough research has been done about the effect of analgesics in treating acute primary headache attacks among children.

Study objective-This study's goal is to describe which medications are used for relieving primary headache attacks in outpatient pediatric population in Israel, and to evaluate their analgesic effect.

Methods: The study group will include 50 patients who were assessed in the pediatric neurology clinic and were diagnosed as having a primary headache.

Evaluation of the results via filled out surveys;

1. First survey for headache assessment at the pediatric neurology clinic.
2. Second survey for tracking given analgesic and its effect by the child at home in addition to checkup calls by pediatric staff.

The survey will include; demographic data, headache diagnosis, baseline headache intensity, antipyretic used and pain assessment.

Research topic:

Use of Common Analgesics in Primary Headaches among Children and Adolescents.

Scientific background:

Headaches are a common complaint in children and adolescents; (1) most cases are caused by a benign problem or a primary headache disorder. Migraine and tension-type headache are the two most common recurring headache patterns seen in children and are distinguished clinically by their characteristics and accompanying features according to the IHS criteria (2).

Treatment of Migraine Frequent Migraine headaches can cause a significant impact on disability, as well as quality of life, prompting the need for early recognition and treatment (3,4,5,6). Thus, the goal of acute treatment of migraine headaches should be a consistent of rapid treatment with minimum side effects and a rapid return to normal function. The most commonly used analgesics are Ibuprofen, and Acetaminophen, and Dipyrone which have shown safety in controlled trials (7). The patient should be instructed to treat the headache as quickly as possible, or at the onset of the aura, if present. Along with treating the acute headache attack, support therapies should be offered by the pediatric neurologist, pediatrician, psychologist, and support groups to reduce the frequency of the attacks.

Acetaminophen and Ibuprofen Efficacy of drugs for the acute treatment of migraine in children has not been studied in well controlled trials. A double-blind crossover study of 88 children was conducted to evaluate the efficacy of Acetaminophen and Ibuprofen, both drugs were shown to be effective and economical treatments for severe to moderate migraine attacks in children. Ibuprofen gave the best relief (8). A similar study was performed on a group of younger children using ibuprofen versus placebo with a similar outcome, although there was a slight male-to-female difference (9).

Dipyrone Dipyrone is used to treat headaches in many countries including Israel. However, it is not available in others, particularly the USA, because of its association with potentially life threatening blood dyscrasias. Its efficacy for the acute treatment of primary headaches in children has not been studied in well controlled trials. Evidence from a small number of trials suggests that Dipyrone is effective for episodic tension-type headache and migraine. No serious adverse events were observed in the included trials, but agranulocytosis is rare and would probably not be observed in such a relatively small sample (10).

In Israel, yet no studies have been initiated to check the efficacy of acute treatment of primary headache attacks among children.

Treatment of TTH Tension type headaches (TTH) are a heterogeneous syndrome, which is diagnosed mainly by the absence of features that are found in other headache types, such as migraine (11). TTH receives much less attention than other types of headache from health authorities, clinical researchers, or industrial pharmacologists. One of the reasons for that may be the fact that most people with infrequent TTH do not consult a doctor for pain relief. They usually manage it themselves using over-the-counter analgesics (12). However, chronic TTH, defined as headache that occurs on 15 days or more per month, is a major health problem with significant educational and socioeconomic effects.

In the case of an acute episode of TTH a gradual strategy is appropriate, as the patients' activity is usually not interrupted and pain intensity is usually not severe (13). In case of repeated, prolonged, or severe episodes of both types of primary headaches, the use of prophylactic treatment should be considered. Pharmacological prophylaxis Life style changes are recommended for young people (1).

Medication overused headaches Medication-overuse headache (MOH) is a chronic headache disorder defined by the International Headache Society as a headache induced by the overuse of analgesics, triptans, or other acute headache compounds. The population-based prevalence of MOH is 0·7% to 1·7%. Most patients with MOH have migraine as their primary headache and overuse triptans or simple analgesics. The pathophysiology of MOH is still unknown. As well as psychological mechanisms such as operant conditioning, changes in endocrinological homoeostasis and neurophysiological changes have been observed in patients with MOH. Recently, a genetic susceptibility has been postulated. In most cases, treatment of MOH consists of abrupt withdrawal therapy and then initiation of an appropriate preventive drug therapy (14).

Purpose of study:

Our goal is to describe which medications are used for relieving primary headache attack in outpatient pediatric population in Israel, and to evaluate their analgesic effect.

Patients and Methods:

The study group will include 50 children 5-18 years of age who were evaluated in the pediatric neurology clinic and were diagnosed as having either migraine or tension type headache. After signing an informed consent the children and/or their parents will be asked to fill a survey about the used of analgesic during acute headache attack, both when they are at the clinic and at home during the headache attack. The surveys will be filled out for a period of 3 months at the first 3 headache episodes. A checkup call by pediatric staff will be performed a month and a half after study initiation, the checkup call's purpose is to make sure the surveys are filled out correctly, follow up and to give medical consultancy when needed. The survey will include; demographic data, headache diagnosis, baseline headache intensity, antipyretic used, dosage, pain assessment at one, three and six-hour time point, migraine-associated symptoms quantification before treatment and at one, three and six-hour time point.

Statistical analysis:

Two-sample t-tests will be performed for continuous variables (headache intensity and treatment) and χ2 for categorical data (such as gender, headache diagnosis). Odds ratios with 95% confidence intervals were computed.

ELIGIBILITY:
Inclusion Criteria:

children 6-18 years of age with migraine headaches. Need for headache abortive treatment -

Exclusion Criteria:

Secondary headache Systemic disease Mental Retardation

-

Ages: 6 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children 6-18 years of age who were diagnosed with migraine headaches will be enrolled into the study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-09-03 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Migraine treatment | 2 hours
  improvement of headache severity

CONTACTS AND LOCATIONS:
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel